CLINICAL TRIAL: NCT05650307
Title: Cardiovascular Imaging to Assess Responses to Metabolic Interventions
Brief Title: CV Imaging of Metabolic Interventions
Acronym: CIRCMeta
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Christopher Nguyen, Director of Cardiovascular Innovation Research Center, The Cleveland Clinic
Other Study IDs: 22-695
Record Dates: First submitted 2022-11-27; First posted 2022-12-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate; Heart Failure; Cardiovascular Diseases
Keywords: MRI; Exercise; Weight loss; Cardiac Rehabilitation; Bariatric Surgery
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Motor Activity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls
  Interventions: Diagnostic Test: MRI
- Bariatric Surgery patients
  Interventions: Diagnostic Test: MRI
- Cardiac rehabilitation patients
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — The magnetic field exposure for MRI in this study is similar to standard clinical MR procedures. The powers of all radio frequency fields in this study are at or under FDA guidelines. The CMR techniques performed here have been used in the literature and in our own clinical cardiac MRI service extensively for several years and have an excellent safety profile in our institution.

SUMMARY:
Cardiovascular disease is the leading cause of death worldwide. It is becoming clearer that heart failure (HF) is closely associated with body's metabolism. Even before the heart becomes weaker, it responds to the stresses by changing the fuels it burns, which results in a reduction in the heart's metabolic efficiency that worsens the heart's condition. Since the heart burns so much fuel and consumes fats and carbohydrates along with other available substrates, any changes in its metabolic efficiency could impact metabolism throughout the body. Specifically, HF is characterized by limited flexibility in substrate utilization leading to an overall energetic deficit. Such energetic deficit is associated with progressive remodeling and alter cardiac hemodynamics. For example, obesity is a widely known risk factor for cardiovascular disease likely lie in how the heart handles energy (substrate utilization and energetics). One commonly recommended treatment for cardiovascular disease, especially coronary artery disease (CAD) or congestive heart failure (CHF), is cardiac rehabilitation. Cardiac rehabilitation for symptomatic cardiovascular disease has been shown to promote a healthy lifestyle, improve physical health and reduce cardiovascular death iii with an apparent dose-dependent response. Participation results in a reduced risk of hospitalization and revascularization procedures, and improved functional status in randomized controlled trials. Thus, cardiac rehabilitation is recommended for individuals with symptomatic CAD or CHF by the American College of Cardiology and American Heart Association. In addition, exercise training in preclinical animal models mirroring the exercise component of cardiac rehabilitation routines have shown increased myocardial regeneration and cardioprotective molecular effects ameliorating adverse myocardial remodeling. Despite these benefits, there is vast heterogeneity in the efficiency of cardiac rehabilitation on the individual level with large variances in improved exercise capacity and cardiac function recovery. Personalization of cardiac rehabilitation necessitates a non-invasive approach to monitor the direct beneficial effects on the heart and more ideally, predict efficacy at baseline. Taken together, understanding how metabolic interventions including bariatric surgery and cardiac rehabilitation change myocardial structure and function is critical for the prevention, diagnosis and prognosis for patients with cardiovascular diseases.

Advanced cardiovascular imaging using Magnetic Resonance Imaging (MRI) has proven to be effective in providing gold standard myocardial tissue characterization. Our team has developed novel cardiac MRI techniques that leverages endogenous tissue properties to reveal a milieu of deep tissue phenotypes including myocardial inflammation, fibrosis, metabolism, and microstructural defects. Among these phenotypes, myocardial microstructure has proven to be most sensitive to early myocardial tissue damage and is predictive of myocardial regeneration. In collaboration with cardiologists at Cleveland Clinic, the investigators aim to study how myocardial microstructure revealed by cardiac MRI changes cardiovascular disease patient population before and after metabolic interventions.

DETAILED DESCRIPTION:
The primary clinical objective of the clinical study is to (1) determine cardiac microstructural phenotypes by cardiac MRI in patients before and after cardiac rehabilitation, or bariatric surgery, and their relationship to cardiac structure/function.

Aim 1: How does the heart's microstructure change before and after cardiac rehabilitation or bariatric surgery? Is this linked to other prevalent macro structure and functional abnormalities and how they change after each metabolic intervention (e.g., cardiac mass or strain)?

Our hypothesis is that characteristic alterations in myocardial microstructure reflected in non-contrast MRI are prevalent in symptomatic cardiovascular disease before and after the respective interventions and may help early detection of cardiovascular disease.

The investigators have chosen a prospective longitudinal cohort design to test the hypothesis that cardiac structure and function change significantly following cardiac rehabilitation or bariatric surgery.

There are TWO arms of the study:

The study protocol for those undergoing cardiac rehabilitation will involve:

* Consent
* MRI at the beginning of 12 weeks of cardiac rehabilitation at Cleveland Clinic. Subjects may opt to complete an MRI of the leg in addition to the cardiac MRI. Patients who opt for both have the option to complete the scans at separate visits.
* Subjects will be scheduled for a 6 week scan if available; however, participation will be optional
* MRI after 12 weeks of cardiac rehabilitation at the Cardiovascular Disease Prevention Center at Cleveland Clinic. If subjects opted to complete both a cardiac scan and a leg scan, the patients have the option to complete these at separate visits.

The study protocol for those who participate in bariatric surgery study:

* Consent
* MRI prior to the bariatric surgery.
* MRI within 12 months of surgery.

Optionally, if the subjects agree, the blood samples will be collected:

• Give blood sample for research purpose only. The blood draw is used to correlate the clinical blood biomarkers to the cardiac MRI data to help us better understand and validate the clinical utility of the novel cardiac MRI techniques. The blood draws should approximately take 20 minutes. The blood draw will take place in the doctor's office or at Mellen center private preparation by a registered nurse or approved technician. The blood will be stored at Lerner freezers until needed for analysis and being analyzed for biomarkers only for this study. It will not be used for future research in the Cleveland Clinic. Only members of the research team will have access to the samples.

The study protocol for healthy volunteers will involve:

* Consent
* One MRI Scan

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Provision of written informed consent
* For bariatric surgery group, obesity (BMI>/=30 kg/m2) and non-obese (BMI <30 kg/m2; for control group)
* For cardiac rehabilitation group, symptomatic cardiovascular disease for patients and no signs of cardiovascular disease for healthy controls

Exclusion Criteria:

* Vulnerable populations will be excluded from this study including Prisoners
* Contraindication to CMR imaging to be determined by standard MRI protocols
* Decisionally impaired (e.g. dementia or cognitive disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 150 subjects (50 for each study arm and 50 healthy controls) will be recruited from the Cleveland Clinic who have been diagnosed with cardiovascular disease and are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2027-09-09 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
Change of Microstructure from baseline and 6-12months | 5 years
  The primary clinical objective of the clinical study is to (1) determine cardiac microstructural phenotypes by cardiac MRI in patients before and after cardiac rehabilitation, or bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Innovation Research Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No